CLINICAL TRIAL: NCT04059848
Title: Transcranial Direct Current Stimulation Combined Neuromuscular Electrical Stimulation on Motor Recovery in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KMUHIRB F(I)-20150053
Record Dates: First submitted 2019-08-14; First posted 2019-08-16 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Chronic Stroke
Keywords: Transcranial direct current stimulation; Neuromuscular electrical stimulation; Stroke; Rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- tDCS combined with NMES (Experimental): In addition to conventional rehabilitation, all subjects received an additional tDCS combined with NMES protocol with a total of 15 sessions for 3 weeks (5 times per week, 30 minutes daily).
  Interventions: Combination Product: tDCS(Intelect Mobile Stimulation and Combination, DJO, France); Combination Product: NMES(Enraf Nonius, Endomed-182, Netherlands)
- tDCS combined with sham NMES (Active Comparator): In addition to conventional rehabilitation, all subjects received an additional tDCS combined with sham NMES protocol with a total of 15 sessions for 3 weeks (5 times per week, 30 minutes daily).
  Interventions: Combination Product: tDCS(Intelect Mobile Stimulation and Combination, DJO, France); Combination Product: NMES(Enraf Nonius, Endomed-182, Netherlands)
- sham tDCS combined with sham NMES (Sham Comparator): In addition to conventional rehabilitation, all subjects received an additional sham tDCS combined with sham NMES protocol with a total of 15 sessions for 3 weeks (5 times per week, 30 minutes daily).
  Interventions: Combination Product: tDCS(Intelect Mobile Stimulation and Combination, DJO, France); Combination Product: NMES(Enraf Nonius, Endomed-182, Netherlands)

INTERVENTIONS:
Combination Product: tDCS(Intelect Mobile Stimulation and Combination, DJO, France)
Combination Product: NMES(Enraf Nonius, Endomed-182, Netherlands)

SUMMARY:
The purpose of this study was to investigate the effects of the combination treatment strategy. A randomized, double-blinded and sham-stimulation study was conducted. Twenty-six participants with chronic stroke (onset > 6 months) were assigned into one of three groups (tDCS combined with NMES, tDCS combined with sham NMES, or sham tDCS combined with sham NMES) by block randomization. In addition to conventional rehabilitation, all subjects received an additional protocol with a total of 15 sessions for 3 weeks (5 times per week, 30 minutes daily). The UE subscale of Fugl-Meyer assessment (UE-FMA) and Action Research Arm Test (ARAT) as primary outcome measures were assessed at beginning of the intervention, after 3-week of treatment, and one-month follow-up. No significant differences in the primary outcome measures at post-treatment and one-month follow-up were found among the tDCS combined with NMES group (n=9), tDCS combined with sham NMES group (n=9), and the sham tDCS combined with sham NMES group (n=8). However, significant changes in UE-FMA (from baseline to post-treatment, p= .02) and ARAT (from baseline to post-treatment, p= .04) score were found for the tDCS combined with NMES group. This preliminary study reveals that the tDCS combined with NMES appears to be beneficial to UE motor recovery after stroke but is not superior to the tDCS alone.

DETAILED DESCRIPTION:
Background and objectives: Previous studies have shown that transcranial direct current stimulation (tDCS) and Neuromuscular electrical stimulation (NMES) could be effective for promoting motor recovery of stroke patients. However, the effects of tDCS combined with NMES on upper extremity (UE) motor recovery in patients with stroke have not been investigated. The purpose of this study was to investigate the effects of the combination treatment strategy. Methods: A randomized, double-blinded and sham-stimulation study was conducted. Twenty-six participants with chronic stroke (onset > 6 months) were assigned into one of three groups (tDCS combined with NMES, tDCS combined with sham NMES, or sham tDCS combined with sham NMES) by block randomization. In addition to conventional rehabilitation, all subjects received an additional protocol with a total of 15 sessions for 3 weeks (5 times per week, 30 minutes daily). The UE subscale of Fugl-Meyer assessment (UE-FMA) and Action Research Arm Test (ARAT) as primary outcome measures were assessed at beginning of the intervention, after 3-week of treatment, and one-month follow-up. Results: Most of the participants had mild to moderate disability in activity of daily living. No significant differences in the primary outcome measures at post-treatment and one-month follow-up were found among the tDCS combined with NMES group (n=9), tDCS combined with sham NMES group (n=9), and the sham tDCS combined with sham NMES group (n=8). However, significant changes in UE-FMA (from baseline to post-treatment, p= .02) and ARAT (from baseline to post-treatment, p= .04) score were found for the tDCS combined with NMES group. Conclusion: This preliminary study reveals that the tDCS combined with NMES appears to be beneficial to UE motor recovery after stroke but is not superior to the tDCS alone.

ELIGIBILITY:
Inclusion Criteria:

* First onset
* Ischemic stroke
* Stroke onset > 6 months
* Brunnstrom recovery stage: ≧3
* Modified Ashworth Scale Elbow flexor : ≦3

Exclusion Criteria:

* Severe language or cognitive impairment
* Orthopaedic or neurological problems
* Pregnancy
* Contraindications for tDCS or NMES

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01-13 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
upper extremity subscale of Fugl-Meyer assessment | at beginning of the intervention, after 3-week of treatment, and one-month follow-up
  The Fugl-Meyer assessment consists of the 33-item upper-extremity (UE-FM) and 17-item lower-extremity subscales.(Fugl-Meyer et al., 1975) The items of the FM are mainly scored on a 3-point scale, from 0 to 2. The total score of the UE-FM ranges from 0 to 66.
Action Research Arm Test | at beginning of the intervention, after 3-week of treatment, and one-month follow-up
  The ARAT(Lyle, 1981) has 19 items in four categories: grasp, grip, pinch, and gross movement. Each item is graded on a 4-point scale, from 0 to 3. The total score has a range of 0 to 57.

IPD SHARING:
Plan to Share IPD: No